CLINICAL TRIAL: NCT02971774
Title: Development of a Multimodal Approach to Assess Stroke Persons Daily Life Activities and Development of a New Tool to Evaluate the Impact of Functional Activites on Quality of Life
Brief Title: Development of a Multimodal Approach to Assess Stroke Patients Daily Life Activities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Sponsor
Other Study IDs: 2005997
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2018-07

CONDITIONS: Stroke in Patients: New Tool to Evaluate the Impact in Their Life
Keywords: stroke; botulinum toxin injection; daily life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- questionnary: self administered questionnary

SUMMARY:
The aim of the study consists in enriching knowledge of health professionals, on the functional difficulties encountered by hemiplegic patients outside the hospital, in particular on hobbies, going out with friends or family, work, daily life and the personal projects. Another objective is to evaluate the diversity of the attitudes and representations of the patients about their body damage. Lastly, the study seeks to develop a new grid of evaluation of the quality of life of the patients, which determines more fields of the existence significantly impacted by the hemiparesy, from the point of view of the patients. It is a question of improving the therapeutic care of the patients and to determine if various therapeutic approaches (occupational, pharmacological, surgical) have an impact on these various fields. The study will be based on qualitative data (interviews) and quantitative (questionnaires).

DETAILED DESCRIPTION:
1. To conduct the research, a sociologist will collaborate with Doctor Nicolas Roche, the study director. The contribution of a sociologist will offer a viewpoint from outside the medical aspect, which will allow more global identification of the areas of the lives of patients that are affected by hemiparesis. Furthermore, the sociological perspective will seek to demonstrate the social aspects, which have heretofore been explored little or not at all in medical and public health studies, such as, for example, in terms of intimacy or self-image. It must delicately capture the practices, logic of action and though of the patients, by placing them in the social contexts in which they evolve and develop. Therefore, attention will be paid to certain "social determinants" (such as sociocultural setting, age or gender) and certain resources (particularly economic, relational and material), which can have an effect on the ways in which patients perceive and cope with the consequences of their hemiparesis. The role of loved ones (partner, family members, friends) will also be examined, since many sociological works have shown that they are usually on the front line to accompany, shape and manage the effects of the motor impairment.
2. The study will target adults regularly followed in the department of physical medicine and rehabilitation of the Raymond-Poincaré hospital. These individuals must present with hemiparesis secondary to a single, hemispheric cerebrovascular accident, be living at home and be able to move inside and outside of the home.

Patients having several severe cognitive disorders or aphasia will not be interviewed.

The study will include an exploration phase (a corpus of approximatively 30 examinations) and a quantitative component (approximatively 100 questionnaires).

Once the examinations have been completed, the preparation of the questionnaire will be done with the validation of clinical experts. The questionnaire will include approximately 20 items, distributed over several dimensions of patients' lives. The participants' response time to the questionnaire should be in a range from 8 to 12 minutes, in order to facilitate its insertion in the professional practices when the patients are at a hospital visit.

The researcher will be in charge of completion of the questionnaire. This will be performed around or during the consultation of patients at Raymond-Poincaré hospital. The first completions will be recorded (with the written approval of surveyed patients) in order to be able to work on possible improvements, particularly in terms of the order of questions or in their understanding and response options. After ten completions, the questionnaire will be slightly revised if modifications appear necessary, then will remain the same until the desired volume of questionnaires is received (approximatively 100).

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* patient with hemiparesis secondary to a single hemispheric cerebrovascular accident
* be living at home
* be able to move inside and outside of the home

Exclusion Criteria:

* Patients having several severe cognitive disorders
* Patients having severe aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will target adults regularly followed in the department of physical medicine and rehabilitation of the Raymond-Poincaré hospital. These individuals must present with hemiparesis secondary to a single, hemispheric cerebrovascular accident, be living at home and be able to move inside and outside of the home.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
daily life questionnary | 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas ROCHE, MD PhD, Principal Investigator — Raymond Poincare Hospital
Locations (1):
- Raymond Poincaré Hospital, Garches, France

IPD SHARING:
Plan to Share IPD: No